CLINICAL TRIAL: NCT00580151
Title: The Use of Clonidine in Pain and Anxiety Associated With Acute Burn Injury in Children
Acronym: clonidine
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Closed due to no response from PI to IRB
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04-101; IFFA (Other: International Firefighters Association)
Record Dates: First submitted 2007-12-18; First posted 2007-12-24 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Pain; Anxiety
Keywords: Pain not controled by morphine; Anxiety not controled by lorazepam
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Clonidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: clonidine
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: clonidine — 3-5 microgram per kilogram every 6 hours for 10 days
  Arms: 1
Drug: placebo — 1 dose every 6 hours
  Arms: 2

SUMMARY:
Some of the children who suffer acute burn injury do not have adequate pain and anxiety management with the current regimen of scheduled opiates (morphine) and benzodiazepines (lorazepam). Other children have significant side effects or contraindications, such as constipation or over sedation, when taking these medications. Clonidine is known to reduce the need for morphine in the management of postoperative pain. The addition of clonidine to the pharmacological treatment of burn wound pain offers a possible adjunct to the standard opiate and benzodiazepines regimen. Clonidine has been used in children in both on a short-term basis (such as postoperative pain management) and on a long-term basis (such as the treatment of attention deficit hyperactivity disorder (ADHD)). This study tests the hypothesis that clonidine in a dose of 5 ug/kilo every 8 hours will be a useful adjunct to the management of pain and anxiety in the acutely burned child. All children will be treated by protocol with morphine (0.03mg/kilo) q4hr prn pain and lorazepam (0.03 mg/kilo) q 4 hours prn anxiety. In addition, after informed consent is obtained the children will be randomized to the addition clonidine or placebo. Pain and anxiety will be assessed using standard instruments blind to the medication being used on a daily basis Also the total dose of morphine and lorazepam during the 10 days of added clonidine or placebo will be recorded.. The pain rating, anxiety ratings, total morphine dose, and total lorazepam dose will be compared between the placebo and clonidine groups with a Student's t test. Once the blind is broken the child will be allowed to remain on the clonidine if it is beneficial. The second year of the grant will expand the age groups down to younger children and also begin to gain information about the effect of clonidine on the hypermetabolic state secondary to burn injury.

ELIGIBILITY:
Inclusion Criteria:

* Pain not controled by morphine
* Anxiety not controled by lorazepam
* Burn injuries of 20% or greater
* Burn type: scald or flame

Exclusion Criteria:

* Small burn injury
* Electrical burns

Ages: 4 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2004-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter J. Meyer III, MD, Principal Investigator — The University of Texas Medical Branch at Galveston
Locations (1):
- Shriners Hospital for Children; Shriners Burns Hospital, Galveston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited in the medical clinic. Recruitment occured between 11/10/04-7/16/05.
Pre-assignment Details: All participants were eligible to participate in the study.
Groups:
- Experimental Group: clonidine : 3-5 microgram per kilogram every 6 hours for 10 days
- Control Group: placebo : 1 dose every 6 hours
Period: Overall Study
Arm/Group | Experimental Group | Control Group
Started | 9 | 0
Completed | 9 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Control Group | Total
Number analyzed (Participants) | 9 | 0 | 9
Age, Categorical [Number; unit: participants]
  <=18 years | 9 |  | 9
  Between 18 and 65 years | 0 |  | 0
  >=65 years | 0 |  | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.8 (3.2) |  | 7.8 (3.2)
Gender [Number; unit: participants]
  Female | 1 |  | 1
  Male | 8 |  | 8
Region of Enrollment [Number; unit: participants]
  United States | 9 |  | 9

OUTCOME MEASURES:

1. Primary Outcome: Pain Reduction
Description: The scale name is "FACES" (Faces Pain Rating Scale). Subjects were asked "rate your WORST PAIN today" (0 = no pain at all, 1-4 = mild pain, 5-6 = moderate pain, 7-9 = severe pain, 10 = excruciating pain). The Faces Pain Rating Scale should be collected every day and then averaged.
Time Frame: Average of the 10 days
Population: Determined by the number of patients recruited.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 9 | 0
units on a scale | .73 [0 to 4] |

2. Secondary Outcome: Anxiety Reduction
Description: The "Fear Thermometer" measures how much fear subject is currently having. (0=None, 1= A little bit, 2= Some, 3= A lot, 4= Very, very much). The average of daily Value for 10 days.
Time Frame: Average of the 10 days
Population: Patients analyzed were all patients consented.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 9 | 0
units on a scale | .76 [0 to 4] |

ADVERSE EVENTS:
Arm/Group | Experimental Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/0
Other Adverse Events (participants affected / at risk) | 0/9 | 0/0

LIMITATIONS AND CAVEATS:
No Adverse Events Recorded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes